CLINICAL TRIAL: NCT03085940
Title: Role of Hydroxychloroquine to Improve Endothelial Dysfunction in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Rudy Hidayat, MD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCQ-ED01
Record Dates: First submitted 2017-02-07; First posted 2017-03-21 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (Experimental)
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine 400mg once daily initially
  Other Names: HCQ
  Arms: Hydroxychloroquine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Rheumatoid arthritis (RA) increase cardiovascular risk and endothelial dysfunction. Hydroxychloroquine (HCQ) is expected to improve endothelial dysfunction through some metabolic effects. The investigators intend to find the role of HCQ to improve endothelial dysfunction in RA patients. This study will also evaluate correlation HOMA-IR (homeostasis model assessment-estimated insulin resistance), FFA (free fatty acid) and ox-LDL (oxidized-LDL) level change, with endothelial dysfunction improvement.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid Arthritis patients (2010 ACR/EULAR criteria)
* Being or will be treated with methotrexate (monotherapy)
* Agree to join the study

Exclusion Criteria:

* Autoimmune diseases other than RA
* Acute severe infection, acute coronary syndrome, heart failure, stroke
* Malignancy or chronic inflammatory diseases
* Eye disease involving the retina and visual field defects
* G6PD (glucose 6-phosphate dehydrogenase) deficiency
* History of smoking within last 5 years
* Lipid lowering, insulin resistance lowering, antidiabetic, insulin, ACE(angiotensin converting enzyme)-inhibitor or ARB(angiotensin receptor blocker) drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Endothelial dysfunction marker | 3 months
  VCAM
Endothelial dysfunction marker | 3 months
  E-Selektine

CONTACTS AND LOCATIONS:
Locations (1):
- Ciptomangunkusumo Hospital, Jakarta, Indonesia